CLINICAL TRIAL: NCT05519085
Title: A Phase 3, Two-Stage, Randomized, Multicenter, Open-Label Study Comparing Mezigdomide (CC-92480), Bortezomib and Dexamethasone (MEZIVd) Versus Pomalidomide, Bortezomib and Dexamethasone (PVd) in Subjects With Relapsed or Refractory Multiple Myeloma (RRMM): SUCCESSOR-1
Brief Title: A Study to Evaluate Mezigdomide, Bortezomib and Dexamethasone (MEZIVd) Versus Pomalidomide, Bortezomib and Dexamethasone (PVd) in Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Acronym: SUCCESSOR-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA057-001; 2023-509859-13 (Other: EU CTR)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Multiple myeloma; RRMM; MeziVd; PVd; CC92480; pomalidomide; bortezomib; dexamethasone; mezigdomide
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MeziVd (mezigdomide, bortezomib and dexamethasone) (Experimental)
  Interventions: Drug: mezigdomide; Drug: Bortezomib; Drug: Dexamethasone
- PVd (pomalidomide, bortezomib and dexamethasone) (Experimental)
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480
  Arms: MeziVd (mezigdomide, bortezomib and dexamethasone)
Drug: Pomalidomide — Specified dose on specified days
  Other Names: Pomalyst; Imnovid; Pom
  Arms: PVd (pomalidomide, bortezomib and dexamethasone)
Drug: Bortezomib — Specified dose on specified days
  Other Names: Velcade; BTZ
Drug: Dexamethasone — Specified dose on specified days
  Other Names: Decadron; Dex

SUMMARY:
The purpose of this study is to compare the efficacy and safety of mezigdomide (CC-92480), bortezomib and dexamethasone (MeziVd) versus pomalidomide, bortezomib and dexamethasone (PVd) in participants with relapsed or refractory multiple myeloma (RRMM) who received between 1 to 3 prior lines of therapy and who have had prior lenalidomide exposure.

ELIGIBILITY:
Inclusion Criteria

- Participant has documented diagnosis of MM and measurable disease, defined as any of the following:.

i) M-protein ≥ 0.5 grams per deciliter (g/dL) by serum protein electrophoresis (sPEP) or.

ii) M-protein ≥ 200 milligrams (mg) per 24-hour urine collection by urine protein electrophoresis (uPEP).

iii) For participants without measurable disease in sPEP or uPEP: serum free light chain (sFLC) levels > 100 mg/L (10 mg/dL) involved light chain and an abnormal kappa/lambda FLC ratio.

* Participants received 1 to 3 prior lines of antimyeloma therapy.
* Participants achieved minimal response [MR] or better to at least 1 prior antimyeloma therapy.

Exclusion Criteria

- Participant has had progression during treatment or within 60 days of the last dose of a proteasome inhibitor, except as noted below:.

i) Subjects who progressed while being treated with, or within 60 days of last dose of bortezomib maintenance given once every 2 weeks (or less frequently) are not excluded.

ii) Participants who progressed while being treated with ixazomib monotherapy maintenance ≥ 6 months prior to the time of starting study treatment are not excluded.

* For participants with prior treatment of a bortezomib containing regimen, the best response achieved was not a minimal response (MR) or better, or participant discontinued bortezomib due to toxicity.
* Participant has had prior treatment with mezigdomide or pomalidomide.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From date of randomization to date of disease progression or death due to any cause (Up to approximately 5 years)

SECONDARY OUTCOMES:
Recommended mezigdomide dose | Up to 12 Months
  Stage 1 only
Plasma concentrations of mezigdomide | Up to 134 Days
  Stage 1 only
Overall Survival (OS) | From date of randomization to date of death due to any cause (Up to approximately 5 years)
Overall Response (OR) | Up to approximately 5 years
  OR is defined as the number of participants who achieve best response of partial response (PR) or better according to the International Myeloma Working Group (IMWG) Response Criteria for Multiple Myeloma
Complete Response (CR) or better | Up to approximately 5 Years
  Defined as the number of participants who achieve best response of complete response (CR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma
Very Good Partial Response (VGPR) or better | Up to approximately 5 years
  Defined as the number of participants who achieve best response of very good partial response (VGPR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma
Time to Response (TTR) | Up to approximately 5 years
Duration of Response (DOR) | Up to approximately 5 years
Time to Progression (TTP) | Up to approximately 5 years
Time to Next Treatment (TTNT) | Up to approximately 5 years
Progression-free Survival 2 (PFS-2) | Up to approximately 5 years
Minimal Residual Disease (MRD) negativity | Up to approximately 5 years
  Defined as the number of participants who achieve complete response (CR) or better and MRD negativity (defined as less than 1 in 10^5 nucleated cells [by next generation flow cytometry] in bone marrow aspirate)
Number of participants with Adverse Events (AEs) | Up to approximately 5 years
Change from baseline in European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC QLQ-C30) scores | Up to approximately 5 years
  The EORTC QLQ-C30 is the most commonly used quality of life instrument in oncology trials. The QLQ-C30 consists of 30 questions incorporated into 5 functional domains physical, role, cognitive, emotional, and social), 9 symptom/other scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a single global Quality of Life (QoL)/global health status score. Items in the functional and symptom scale use raw participant response of 1 to 4, where 1 = "not at all" and 4 = "very much." The 2 global items contain responses ranging from 1 "very poor" to 7 "excellent." The recall period is 1 week. All domain scores are transformed in a range from 0 to 100, where a higher functional score indicates more favorable outcomes and a higher score on the symptom domains indicates a less favorable participant outcome. Stage 2 only.
Change from baseline in European Organization for Research and Treatment of Cancer - Quality of Life Multiple Myeloma Module (EORTC QLQ-MY20) score | Up to approximately 5 years
  The EORTC QLQ-MY20 is a 20-item myeloma module intended for use among participants varying in disease stage and treatment modality. Participants rate symptoms or problems on a scale from 1 to 4 where 1 = "not at all" and 4 = "very much." Stage 2 only.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (266):
- United States (56):
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Sharp Memorial Hospital, San Diego, California
  - Local Institution - 0273, West Hollywood, California
  - Local Institution - 0381, Aurora, Colorado
  - UConn Health, Farmington, Connecticut
  - Local Institution - 0208, New Haven, Connecticut
  - Advanced Research, Coral Springs, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - University Cancer Blood Ctr, Athens, Georgia
  - Local Institution - 0048, Marietta, Georgia
  - Local Institution - 0330, Garden City, Kansas
  - University of Kansas Medical Center, Westwood, Kansas
  - Our Lady of the Lake RMC, Baton Rouge, Louisiana
  - Local Institution - 0255, New Orleans, Louisiana
  - Local Institution - 0385, Shreveport, Louisiana
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Local Institution - 0242, Jackson, Mississippi
  - Astera Cancer Care, East Brunswick, New Jersey
  - Local Institution - 0363, Ridgewood, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Local Institution - 0245, Buffalo, New York
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Local Institution - 0373, New Hyde Park, New York
  - Local Institution - 0371, New York, New York
  - Rochester General Hospital, Rochester, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Local Institution - 0372, The Bronx, New York
  - Local Institution - 0274, Williamsville, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital, Mayfield Heights, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Local Institution - 0264, York, Pennsylvania
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Texas Oncology - West Texas, Abilene, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - VA Puget Sound Health Care System, Seattle, Washington
  - Local Institution - 0293, Seattle, Washington
  - Local Institution - 0097, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Local Institution - 0220, Madison, Wisconsin
- Argentina (7):
  - Sanatorio Chivilcoy, Chivilcoy, Buenos Aires
  - Centro Medico Barrio Parque, Buenos Aires, Buenos Aires F.D.
  - Hospital Privado Universitario de Córdoba, Córdoba, Córdoba Province
  - Clinica Viedma S. A, Viedma, R
  - Hospital Privado de Rosario, Rosario, Santa Fe Province
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, S3000epv, Santa Fe Province
  - Hospital Británico de Buenos Aires, Buenos Aires
- Australia (8):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Wollongong Hospital-Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (5):
  - Klinik Ottakring, Vienna, Vienna
  - Universitätsklinikum Krems, Krems
  - LKH Hochsteiermark - Standort Leoben, Leoben
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Hanusch-Krankenhaus, Vienna
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Campus St.-Jan, Genk, Limburg
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - ZNA Cadix, Antwerp
- Brazil (7):
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador, Estado de Bahia
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia e Oncologia, Joinville, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Americas Centro de Oncologia Integrado, Rio de Janeiro
  - Clínica Médica São Germano S/S Ltda, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (3):
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre, Greenfield Park, Quebec
  - Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal (CIUSSS NÎM) - Hôpital du Sacré-Coeur, Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
- Chile (3):
  - Centro de Investigaciones, Viña del Mar, Región de Valparaíso
  - Clínica Inmunocel, Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (36):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Local Institution - 0165, Beijing, Beijing Municipality
  - Local Institution - 0141, Beijing, Beijing Municipality
  - The First Afffiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - Henan Cancer Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Local Institution - 0168, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital - Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - Guangxi Medical University No.1 Affiliated Hospital, Nanning, Guangxi
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - People's Hospital of Henan Province, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University Respiratory, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Local Institution - 0110, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai 6th people's hospital, Shanghai, Shanghai Municipality
  - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Local Institution - 0356, Deyang, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Local Institution - 0353, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Local Institution - 0151, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Shanxi Bethune Hospital;Shanxi Academy of Medical Sciences, Taiyuan
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (2):
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki
- France (10):
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg, Alsace
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Centre Leon Berard, Lyon Cedex08, Auvergne-Rhône-Alpes
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Nîmes - Institut de Cancérologie du Gard - Hôpital Universitaire Carémeau, Nîmes
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
  - Hôpital Saint Antoine, Paris, Île-de-France Region
- Germany (16):
  - TUM Klinikum, München, Bavaria
  - Klinikum Traunstein, Traunstein, Bavaria
  - Medizinisches Versorgungszentrum, Weiden, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Praxis Onkologie am Raschplatz, Hanover, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Marien Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Local Institution - 0396, Erfurt, Thuringia
  - Universitätsklinikum Aachen, Aachen
  - Sozialstiftung Bamberg, Bamberg
  - Gemeinschaftspraxis Hämatologie - Onkologie Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Altona, Hamburg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Gemeinschaftspraxis Dres. med. Björn Schöttker & Dominik Pretscher, Würzburg
- Greece (3):
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - G. Papanikolaou General Hospital, Thessaloniki, Thessaloníki
- India (8):
  - HCG Aastha Cancer Centre, Ahmedabad, Gujarat
  - Marengo Asia Hospitals Gurugram, Gurugram, Haryana
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi, Karnataka
  - Mumbai Oncocare Centre - Nanachowk, Mumbai, Maharashtra
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - Tata Memorial Centre - Homi Bhabha Cancer Hospital, Varanasi, Uttar Pradesh
  - Christian Medical College & Hospital, Ludhiana
  - Jawaharlal Institute Of Postgraduate Medical Education And Research, Puducherry
- Ireland (4):
  - University College Hospital - Galway, Galway, Connacht
  - Cork University Hospital, Cork
  - St. James's Hospital, Dublin
  - Local Institution - 0251, Limerick
- Israel (6):
  - Meir Medical Center, Kfar Saba, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center - Do Not Use - Duplicate Facility, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, Tall Abīb
  - Rabin Medical Center, Peatch Tikva
- Italy (5):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Azienda Ospedaliera Sant'Andrea, Rome, Roma
  - Policlinico "G. Rodolico", Catania, Sicily
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Japan (18):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Japan Community Healthcare Organization Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Mito Medical Center, Higashiibaraki, Ibaraki
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho, Iwate
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Saitama Medical University Hospital, Iruma, Saitama
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun, Shizuoka
  - Nihon University Itabashi Hospital, Itabashiku, Tokyo
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Kumamoto University, Kumamoto
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - The Jikei University Hospital, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
- New Zealand (4):
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Dunedin Hospital, Dunedin, Otago
  - Auckland City Hospital, Auckland
  - Local Institution - 0334, Auckland
- Poland (6):
  - Local Institution - 0346, Skórzewo, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0325, Krakow, Lesser Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Local Institution - 0292, Słupsk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice
- Portugal (3):
  - Hospital de Braga, Braga
  - Champalimaud Foundation, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Local Institution - 0355, San Juan, Puerto Rico
- Romania (3):
  - Fundeni Clinical Institute, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi, Iași
- South Africa (4):
  - Netcare Pretoria East Hospital, Centurion, GP
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Haemalife, Kuilsriver, Western Cape
  - Constantiaberg Haematology, Plumstead, Western Cape
- South Korea (16):
  - Local Institution - 0106, Busan, Busan
  - Pusan National University Hospital, Busan, Busan
  - Local Institution - 0102, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam, Gyeonggido
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - Local Institution - 0103, Hwasun, Jeonranamdo
  - Local Institution - 0101, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0104, Seoul, Seoul Teugbyeolsi
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0105, Seoul, Seoul-teukbyeolsi
  - Local Institution - 0100, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Local Institution, Seoul
- Spain (10):
  - Local Institution - 0183, Palma, Balearic Islands
  - Hospital Universitari Son Espases, Palma, Balears [Baleares]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0073, Barcelona, Catalunya [Cataluña]
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia, Región de
  - Hospital Costa del Sol, Marbella, Málaga
  - Local Institution - 0182, Marbella, Málaga
  - Hospital San Pedro de Alcantara, Cáceres
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (6):
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Liv Hospital Ankara, Ankara
  - Istanbul University, Istanbul Faculty of Medicine, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Ondokuz Mayıs Universitesi, Samsun
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - The Royal Cornwall Hospital, Truro, England
  - Lanarkshire NHS Trust - Monklands Hospital, Airdrie, Great Britain
  - King's College Hospital, London, Greater London
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Hammersmith Hospital, London, London, City of
  - Barnet Hospital, Barnet
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05519085.html